CLINICAL TRIAL: NCT05729321
Title: Lock sOlutiOnS for Epicutaneo-caval Catheters in Neonates: a "LOOSEN" Pilot Study
Acronym: LOOSEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D ANDREA VITO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4880
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Catheter-related Bloodstream Infection; Preterm; Catheter Infection; Catheter Complications
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epicutaneo-caval catheter removed electively: This is a pilot study designed to evaluate the patency of the Epicutaneo-caval catheter after its closure for 1 hour in order to assess the feasibility of possible Taurolidine lock-terapy in Epicutaneo-Caval Catheters.
  Interventions: Combination Product: neutrox

INTERVENTIONS:
Combination Product: neutrox — Each ECC, after discontinuing the Parental Nutrition (NP) infusion, will be flushed with 0.3 ml saline. Subsequently, Saline will be infused at a rate of 2 ml/h for 10 minutes. The ECC will then be closed for 1 hour. At the end of the hour the ECC will be once again flushed with 0.3 ml Saline and infused with SF at the rate of 2 cc/h for 10 minutes. The difference in pressure of the two infusions, before and after catheter closure, will be evaluated.

SUMMARY:
Epicutaneo-caval catheters (ECCs) are widely used in neonatal intensive care units (NICUs). They are small catheters inserted via superficial veins of the limbs or scalp using direct vein visualization The pathogenic microorganisms colonized inside catheters can easily form a bacterial biofilm and eventually spread with blood flow which causes bloodstream infection. Many authors have studied the antibiotic-lock therapy (ALT) in which a high-dose antibiotic solution is dripped and maintained in the catheter cavity for a certain period and can dissolve the biofilm formed on the wall to reduce the colonization of the bacteria and kill the embedded bacteria.The aim of the study is to evaluate the patency of the Epicutaneo-caval catheter after its closure for 1 hour.

ELIGIBILITY:
Inclusion Criteria:

All the Epicutaneo-caval catheter that need to be removed electively will be included in the study -

Exclusion Criteria:

All the Epicutaneo-caval catheters removed not electively but for infectious or mechanical complications will be excluded from the study.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All infants who have catheters that need to be removed electively.
Sampling Method: Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Pressure level mmHg | 1 hours
  The aim of the study is to evaluate the patency of the Epicutaneo-caval catheter after its closure for 1 hour.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Fondazione Policlinico Gemelli IRCSS, Roma, Itsly
  - FPGemelliIRCCS, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jain A, Deshpande P, Shah P. Peripherally inserted central catheter tip position and risk of associated complications in neonates. J Perinatol. 2013 Apr;33(4):307-12. doi: 10.1038/jp.2012.112. Epub 2012 Sep 6. PMID 22955288
- [Background] Barone G, Pittiruti M. Epicutaneo-caval catheters in neonates: New insights and new suggestions from the recent literature. J Vasc Access. 2020 Nov;21(6):805-809. doi: 10.1177/1129729819891546. Epub 2019 Dec 5. PMID 31804149
- [Background] Barone G, Pittiruti M, Biasucci DG, Elisei D, Iacobone E, La Greca A, Zito Marinosci G, D'Andrea V. Neo-ECHOTIP: A structured protocol for ultrasound-based tip navigation and tip location during placement of central venous access devices in neonates. J Vasc Access. 2022 Sep;23(5):679-688. doi: 10.1177/11297298211007703. Epub 2021 Apr 5. PMID 33818191
- [Background] Viale P, Pagani L, Petrosillo N, Signorini L, Colombini P, Macri G, Cristini F, Gattuso G, Carosi G; Italian Hospital and HIV Infection Group. Antibiotic lock-technique for the treatment of catheter-related bloodstream infections. J Chemother. 2003 Apr;15(2):152-6. doi: 10.1179/joc.2003.15.2.152. PMID 12797393
- [Background] Dumichen MJ, Seeger K, Lode HN, Kuhl JS, Ebell W, Degenhardt P, Singer M, Geffers C, Querfeld U. Randomized controlled trial of taurolidine citrate versus heparin as catheter lock solution in paediatric patients with haematological malignancies. J Hosp Infect. 2012 Apr;80(4):304-9. doi: 10.1016/j.jhin.2012.01.003. Epub 2012 Feb 18. PMID 22342714